CLINICAL TRIAL: NCT02813993
Title: Couples Fertility and Pregnancy Awareness
Acronym: CFPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FPCEUP/RH2; SFRH/BD/103234/2014 (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia)
Record Dates: First submitted 2016-06-17; First posted 2016-06-27 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2020-03

CONDITIONS: Fertility; Decision to Get Pregnant
Keywords: infertility; fertility awareness; preconceptional care; health interventions; couples
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): A five-minute video concerning age-related fertility decline, fertility risk factors, success of infertility treatments and emotional consequences of childlessness
  Interventions: Other: Health educational video
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Health educational video
  Arms: Intervention Group

SUMMARY:
Recent evidence has shown that young people that want to have children have low fertility knowledge. This study evaluates the efficacy of a video intervention on fertility knowledge, on changes in lifestyle and on the decision to start to get pregnant.

DETAILED DESCRIPTION:
This study will compare the efficacy of a video intervention versus control (no video) in couples that intend to have children in the next three years. The couples will be randomized to the two groups. The video contains information concerning age-related fertility decline, fertility risk factors, the success of infertility treatments, and emotional consequences of childlessness.

ELIGIBILITY:
Inclusion Criteria:

* Female member of the couples has between 24 to 40 years
* Childless couples trying to conceive or couples who desired to have children in the next 3 years
* Relationship length minimum of one year

Exclusion Criteria:

* Couples that already had achieved a successful pregnancy
* Couples with children

Ages: 24 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 244 (Actual)
Dates: Start 2016-10; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Change in Fertility knowledge | T0 - before the intervention; T1 - one month later; T2 - six months later; T3 - one year later
  This measure assesses fertility knowledge by asking questions on the probability of conception and fertility treatment success rates, infertility definition and infertility risk factors

SECONDARY OUTCOMES:
Change in number of months planned to get pregnant/pregnancy | T0 - before the intervention; T1 - one month later; T2 - six months later; T3 - one year later
  This question measures the number of months estimated by participants until they get pregnant or pregnancy
Change in intention and adoption of fertility-optimizing behaviors | T0 - before the intervention; T1 - one month later; T2 - six months later; T3 - one year later
  These questions assessed the intentions to adopt and the effective adoption of fertility-optimizing behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Pedro, MSc, Principal Investigator — Universidade do Porto
Locations (1):
- University of Porto, Faculty of Psychology and Educational and Education Sciences, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided